CLINICAL TRIAL: NCT04390503
Title: A Phase 2 Randomized, Double-blinded Trial to Evaluate the Efficacy and Safety of Human Anti-SARS-CoV-2 Plasma for Early Treatment of COVID-19
Brief Title: Convalescent Plasma for Early Treatment of COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment challenges
Sponsor: Andrew Eisenberger (Other)
Responsible Party: Sponsor-Investigator, Andrew Eisenberger, Associate Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAT0052
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: SARS-CoV 2; COVID-19
Keywords: Coronavirus; COVID; Convalescent Plasma
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: A total of 150 eligible subjects will be randomized in a 2:1 ratio to receive either convalescent plasma qualitatively positive for SARS-CoV-2 antibody (anti-SARS-CoV-2 plasma) or control (albumin 5%)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Convalescent Plasma (anti-SARS-CoV-2 plasma) (Experimental): Participants randomized to the experimental arm will receive 2 units (approximately 200 to 250 mL per unit, total 400-500mL) of convalescent plasma that was collected from a volunteer who recovered from COVID-19 disease.
  Interventions: Biological: Convalescent Plasma (anti-SARS-CoV-2 plasma)
- Control (albumin 5%) (Active Comparator): Participants randomized to the control arm will receive 2 units of 250 mL (500mL total) of albumin (human) 5% infusion. The albumin will be prepared in bags that are identical to the bags used for plasma. The similar appearance of albumin and plasma will facilitate maintaining the blinded status of subjects and most of the study staff.
  Interventions: Biological: Control (albumin 5%)

INTERVENTIONS:
Biological: Convalescent Plasma (anti-SARS-CoV-2 plasma) — Convalescent Plasma that contains antibody titers against SARS-CoV-2.
  Arms: Convalescent Plasma (anti-SARS-CoV-2 plasma)
Biological: Control (albumin 5%) — Albumin (Human) 5% is a sterile aqueous solution for intravenous use containing the albumin component human plasma.
  Arms: Control (albumin 5%)

SUMMARY:
This is a double-blinded, randomized control trial to assess the efficacy and safety of anti-SARS-CoV-2 convalescent plasma as early treatment. Participants will be randomized 2:1 to receive either convalescent plasma qualitatively positive for SARS-CoV-2 antibody ("anti-SARS-CoV-2 plasma") or control (albumin 5%). This study will investigate the potential of convalescent plasma (CP) to reduce severity of and/or help treat SARS-CoV-2 disease in patients with mild disease.

DETAILED DESCRIPTION:
There are no approved therapies for Coronavirus disease 2019 (COVID-19), also known as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Exposure to viruses results in an adaptive immune response that commonly include antibodies with neutralization activity. Plasma from subjects who have recovered from viral infections has been used to both prevent or treat disease. Notable examples of the successful use of convalescent plasma (CP) include influenza, measles, Argentine hemorrhagic fever, Middle East respiratory syndrome (MERS), Ebola and severe acute respiratory syndrome (SARS). In recent work in China, an open label safety trial of CP in patients with COVID-19 suggested a substantive benefit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older
* Recent close contact with a person with COVID-19, i.e. last close contact occurred within 7 days of anticipated infusion of study product. It is anticipated that most contacts will be household contacts with extensive interaction. All must meet the CDC criteria for close contacts. This includes healthcare workers at higher risk of developing severe disease.

OR

* Recent self-reported or documented evidence of infection by nasal swab PCR that is positive for SARS-CoV-2, i.e., nasal sample was collected within 7 days or 10 days of anticipated infusion of study product for those who are asymptomatic or symptomatic, respectively.
* Evidence of infection by nasal swab PCR that is positive for SARS-CoV-2 at screening visit.
* May or may not be hospitalized.
* No symptoms or no more than 5 days of mild symptoms at the time of screening. Mild symptoms (rated by participant as mild and not interfering with normal daily activities) may include:

  * Mild rhinorrhea
  * Mild sore throat or throat irritation
  * Mild nonproductive cough
  * Mild fatigue (able to perform Activities of Daily Living (ADLs))
* Risk for severe COVID-19 based on a risk score of ≥ 1 Calculated Risk Score of ≥ 1 point, with risk factors based on Center for Disease Control and Prevention (CDC) description

  * Age 65-74: 1 point
  * Age ≥ 75: 2 points
  * Known cardiovascular disease (including hypertension): 1 point
  * Diabetes mellitus: 1 point
  * Pulmonary disease (COPD, moderate to severe asthma, current smoking or other): 1 point
  * Morbid obesity: 1 point
  * Immunocompromised state: 1 point Received a bone marrow or solid organ transplant at any time, received chemotherapy for a malignancy within the past 6 months, has an acquired or congenital immunodeficiency, currently receiving immunosuppressive or immune modulating medications, HIV with non-suppressed viral load and/or cluster of differentiation 4 (CD4+) T cell count <200 cells/mL).

Exclusion Criteria:

* Receipt of any blood product in past 120 days.
* Psychiatric or cognitive illness or recreational drug/alcohol use that in the opinion of the principal investigator, would affect subject safety and/or compliance.
* Confirmed or self-reported presumed COVID-19, with symptoms that began more than 5 days prior to enrollment, and SARS-CoV-2 PCR positive sample that was collected more than 7 days prior to anticipated infusion for an asymptomatic participant or more than 10 days prior to anticipated infusion for a patient with mild symptoms at screening.
* Symptoms consistent with COVID---19 infection that are more than mild (as defined above) at time of screening.
* Symptoms consistent with COVID---19 infection that are more than mild at time of screening.
* History of allergic reaction to transfusion blood products
* Inability to complete infusion of the product within 48 hours after randomization.
* Resident of a long term or skilled nursing facility
* Known prior diagnosis of immunoglobulin A (IgA) deficiency
* Oxygen saturation that is < 95% at the screening visit
* On supplemental oxygen at time of enrollment
* Participation in another clinical trial of anti-viral agent(s) for COVID-19
* Receipt of any COVID-19 vaccine, either as part of a clinical research trial or through routine service delivery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Justman, MD, Principal Investigator — Columbia University
Locations (1):
- National Institute of Infectious Diseases Evandro Chagas (INI), Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arabi YM, Hajeer AH, Luke T, Raviprakash K, Balkhy H, Johani S, Al-Dawood A, Al-Qahtani S, Al-Omari A, Al-Hameed F, Hayden FG, Fowler R, Bouchama A, Shindo N, Al-Khairy K, Carson G, Taha Y, Sadat M, Alahmadi M. Feasibility of Using Convalescent Plasma Immunotherapy for MERS-CoV Infection, Saudi Arabia. Emerg Infect Dis. 2016 Sep;22(9):1554-61. doi: 10.3201/eid2209.151164. PMID 27532807
- [Background] Casadevall A, Dadachova E, Pirofski LA. Passive antibody therapy for infectious diseases. Nat Rev Microbiol. 2004 Sep;2(9):695-703. doi: 10.1038/nrmicro974. PMID 15372080
- [Background] Casadevall A, Pirofski LA. Antibody-mediated regulation of cellular immunity and the inflammatory response. Trends Immunol. 2003 Sep;24(9):474-8. doi: 10.1016/s1471-4906(03)00228-x. No abstract available. PMID 12967670
- [Background] Casadevall A, Scharff MD. Serum therapy revisited: animal models of infection and development of passive antibody therapy. Antimicrob Agents Chemother. 1994 Aug;38(8):1695-702. doi: 10.1128/AAC.38.8.1695. No abstract available. PMID 7985997
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Crowe JE Jr, Firestone CY, Murphy BR. Passively acquired antibodies suppress humoral but not cell-mediated immunity in mice immunized with live attenuated respiratory syncytial virus vaccines. J Immunol. 2001 Oct 1;167(7):3910-8. doi: 10.4049/jimmunol.167.7.3910. PMID 11564809
- [Background] Gunn BM, Yu WH, Karim MM, Brannan JM, Herbert AS, Wec AZ, Halfmann PJ, Fusco ML, Schendel SL, Gangavarapu K, Krause T, Qiu X, He S, Das J, Suscovich TJ, Lai J, Chandran K, Zeitlin L, Crowe JE Jr, Lauffenburger D, Kawaoka Y, Kobinger GP, Andersen KG, Dye JM, Saphire EO, Alter G. A Role for Fc Function in Therapeutic Monoclonal Antibody-Mediated Protection against Ebola Virus. Cell Host Microbe. 2018 Aug 8;24(2):221-233.e5. doi: 10.1016/j.chom.2018.07.009. PMID 30092199

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Arm: Convalescent Plasma: Participants will receive 2 units (approximately 200 to 250 mL per unit, total 400-500mL) of convalescent plasma that was collected from a volunteer who recovered from COVID-19 disease.
- Control Arm: Albumin 5%: Participants will receive 2 units of 250 mL (500mL total) of human albumin 5% infusion. Albumin 5% is a sterile aqueous solution for intravenous use containing the albumin component human plasma. The albumin will be prepared in bags that are identical to the bags used for plasma. The similar appearance of albumin and plasma will facilitate maintaining the blinded status of subjects and most of the study staff.
Period: Overall Study
Arm/Group | Experimental Arm: Convalescent Plasma | Control Arm: Albumin 5%
Started | 150 | 73
Completed | 147 | 72
Not Completed | 3 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm: Convalescent Plasma | Control Arm: Albumin 5% | Total
Number analyzed (Participants) | 150 | 73 | 223
Age, Customized [Count of Participants; unit: Participants]
  <60 years | 74 | 28 | 102
  60-69 years | 35 | 24 | 59
  70-79 years | 28 | 16 | 44
  ≥80 years | 13 | 5 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 51 | 147
  Male | 54 | 22 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 101 | 49 | 150
  United States | 49 | 24 | 73
Clinical status at randomization [Count of Participants; unit: Participants]
  Hospitalized, not requiring supplemental oxygen | 5 | 5 | 10
  Hospitalized, requiring supplemental oxygen, HFO, NIV | 125 | 57 | 182
  Hospitalized, requiring IMV, ECMO, or both | 17 | 11 | 28
Baseline conditions [Count of Participants; unit: Participants]
  COVID-19 | 150 | 73 | 223
  Hypertension | 53 | 22 | 75
  Diabetes mellitus | 55 | 27 | 82
  Hyperlipidemia | 27 | 9 | 36
  Chronic cardiac disease | 56 | 28 | 84
  Chronic kidney disease | 13 | 8 | 21
  Chronic pulmonary disease | 15 | 5 | 20
  Chronic liver disease | 3 | 1 | 4
  HIV | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Non-Hospitalized Participants
Description: Participants who were discharged from the hospital after receiving the study intervention.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm: Convalescent Plasma | Control Arm: Albumin 5%
Number analyzed (Participants) | 150 | 73
Participants | 108 | 48

2. Primary Outcome: Number of Hospitalized Participants Requiring Supplemental Oxygen
Description: Participants who remained hospitalized and required supplemental oxygen after receiving the study drug.
Time Frame: Up to 28 days
Population: Only includes individuals who have data at day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm: Convalescent Plasma | Control Arm: Albumin 5%
Number analyzed (Participants) | 42 | 25
Participants | 7 | 1

3. Primary Outcome: Number of Hospitalized Participants Requiring High-flow Oxygen Therapy or Noninvasive Mechanical Ventilation
Description: Participants who remained hospitalized and required high-flow oxygen therapy or noninvasive mechanical ventilation after receiving the study intervention.
Time Frame: Up to 28 days
Population: Only includes individuals who have data at day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm: Convalescent Plasma | Control Arm: Albumin 5%
Number analyzed (Participants) | 42 | 25
Participants | 1 | 0

4. Secondary Outcome: Number of In-hospital Mortalities
Description: Participants who died in the hospital after receiving the study drug.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm: Convalescent Plasma | Control Arm: Albumin 5%
Number analyzed (Participants) | 150 | 73
Participants | 19 | 18

5. Secondary Outcome: Rate of Measurable Anti-SARS-CoV-2 Titers
Description: To compare the rate of measurable anti-SARS-CoV-2 titers between recipients of CP (anti-SARS-CoV-2 plasma) versus control (albumin 5%).
Time Frame: Up to 90 days
Population: These samples were not collected for analysis.
Groups:
- All Participants: Includes all individuals who were consented and randomized.
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Rate of SARS-CoV-2 PCR Positivity
Description: Compare the rates of SARS-CoV-2 PCR positivity (RT PCR) amongst the anti-SARS-CoV-2 convalescent plasma and control (albumin 5%).
Time Frame: Up to 28 days
Population: These samples were not collected for analysis.
Arm/Group | All Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of SARS-CoV-2 PCR Positivity
Description: Compare the duration of SARS-CoV-2 PCR positivity (RT PCR) amongst the anti-SARS-CoV-2 convalescent plasma and control (albumin 5%).
Time Frame: Up to 28 days
Population: Data was not collected for this outcome measure.
Arm/Group | All Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: Levels of SARS-CoV-2 RNA
Description: Compare the levels of SARS-CoV-2 RNA between the recipients of antiSARS-CoV-2 plasma and control (albumin 5%)
Time Frame: Up to 28 days
Population: Samples were not collected for analysis.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Collected from baseline until day 28.
Description: Adverse Events and Serious AEs were only collected from participants who completed the study (i.e., 147 participants in the Experimental Arm and 72 participants in the Control Arm).
Arm/Group | Experimental Arm: Convalescent Plasma | Control Arm: Albumin 5%
All-Cause Mortality (participants affected / at risk) | 19/150 | 18/73
Serious Adverse Events (participants affected / at risk) | 39/147 | 26/72
Other Adverse Events (participants affected / at risk) | 38/147 | 17/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm: Convalescent Plasma (N=147) | Control Arm: Albumin 5% (N=72)
arterial thrombosis (Blood and lymphatic system disorders) | 0 | 1
disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
pulmonary embolism (Blood and lymphatic system disorders) | 2 | 0
venous thrombosis (Blood and lymphatic system disorders) | 4 | 2
arrhythmia (Cardiac disorders) | 10 | 5
cardiac arrest (Cardiac disorders) | 1 | 3
cardiogenic shock (Cardiac disorders) | 0 | 1
myocarditis (Cardiac disorders) | 1 | 0
septic shock (Cardiac disorders) | 4 | 4
pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
hypothermia (Immune system disorders) | 0 | 1
ventilator-associated pneumonia (Infections and infestations) | 2 | 2
ketoacidosis (Renal and urinary disorders) | 1 | 0
metabolic acidosis (Renal and urinary disorders) | 0 | 1
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 24 | 16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm: Convalescent Plasma (N=147) | Control Arm: Albumin 5% (N=72)
diarrhea (Gastrointestinal disorders) | 9 | 3
Pneumonia (Infections and infestations) | 16 | 7
hypotension (Cardiac disorders) | 8 | 6
anemia (Blood and lymphatic system disorders) | 12 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT04390503/Prot_SAP_000.pdf